CLINICAL TRIAL: NCT03095352
Title: A Randomized Phase II Study of Pembrolizumab, an Anti-Programmed Cell Death (PD)-1 Antibody, in Combination With Carboplatin Compared to Carboplatin Alone in Breast Cancer Patients With Chest Wall Disease
Brief Title: Pembrolizumab With Carboplatin Compared to Carboplatin Alone in Breast Cancer Patients With Chest Wall Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laura Huppert, MD, BA (Other)
Collaborators: Mayo Clinic (Other); Johns Hopkins University (Other); Translational Breast Cancer Research Consortium (Other); Massachusetts General Hospital (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Laura Huppert, MD, BA, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC#157521+167513; TBCRC 044 (Other: Translational Breast Cancer Research Consortium); NCI-2018-00010 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-03-24; First posted 2017-03-29 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Chest Wall Disease
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; Carboplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Pembrolizumab + Carboplatin (Experimental): Participants receive carboplatin intravenously (IV) and pembrolizumab IV over 30 minutes on day 1. Participants who are HER2+ also receive trastuzumab IV every 3 weeks. Treatment repeats every 3 weeks for a least 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 cycles of carboplatin and pembrolizumab, participants with stable or responding disease receive pembrolizumab monotherapy on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Biological: Trastuzumab
- Arm B: Carboplatin Monotherapy (Experimental): Participants receive carboplatin on day 1. Patients who are HER2+ also receive trastuzumab IV every 3 weeks. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Participants with disease progression (PD) are eligible to receive pembrolizumab on day 1 of each cycle (crossover). Carboplatin may be continued or added back into the treatment regimen at the investigator's discretion. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Biological: Trastuzumab

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg Given IV
  Other Names: Keytruda
  Arms: Arm A: Pembrolizumab + Carboplatin
Drug: Carboplatin — Arm A: area under the curve (AUC) 5 IV every 3 weeks Arm B: AUC 5 IV every 3 weeks
  Other Names: Ribocarbo
Biological: Trastuzumab — For HER2+ patients: IV every 3 weeks using standard approved dosing
  Other Names: Herceptin

SUMMARY:
This is a phase II multicenter study including breast cancer patients with chest wall disease that is hormone resistant (estrogen receptor (ER) positive/progesterone receptor (PR) positive/human epidermal growth factor receptor 2 (HER2) negative breast cancer with progressive disease on 2 prior lines of hormonal therapy) or triple negative (ER negative/PR negative/HER2 negative, TNBC).

A companion translational study is operating concurrently with the study described above. In this study, biomarker research to be performed on tumor biopsies and peripheral blood samples will be performed to explore the immunologic and genomic mechanism of action underlying treatment with pembrolizumab and carboplatin versus carboplatin alone. This protocol includes tissue and blood correlative exploratory endpoints including changes in tumor PD-L1 (programmed death ligand 1) gene expression, tumor and peripheral blood immune composition and cytokine expression, plasma tumor DNA, circulating tumor cells, and tumor myelocytomatosis (MYC) oncogene expression using tumor biopsy and peripheral blood testing before and after treatment; correlations with these markers and disease control rate will be assessed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the disease control rate (including complete response (CR), partial response (PR) and stable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 at 18 weeks of treatment in breast cancer patients with chest wall disease treated with pembrolizumab and carboplatin or carboplatin alone.

SECONDARY OBJECTIVES:

I. To determine the disease control rate (including CR, PR and stable disease as defined by Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) at 18 weeks of treatment in breast cancer participants with chest wall disease treated with pembrolizumab and carboplatin or carboplatin alone.

II. To determine progression free survival (PFS) in participants treated with pembrolizumab and carboplatin vs. carboplatin alone.

III. To determine the toxicity of pembrolizumab and carboplatin vs. carboplatin alone.

IV. To determine 18 week disease control rate (DCR) based on tumor programmed death-ligand 1 (PD-L1) expression via immunohistochemistry.

V. To determine the overall response rate (ORR) of participants treated with pembrolizumab and carboplatin vs. carboplatin alone.

OUTLINE:

Participants will be enrolled at Translational Breast Cancer Research Consortium (TBCRC) sites and will be randomized 2:1 to receive treatment with pembrolizumab and carboplatin (n=56, Arm A) or carboplatin alone (n=28, Arm B) until documented disease progression.

Participants randomized to Arm B may cross-over after documented disease progression to pembrolizumab with or without carboplatin at investigator's discretion. Participants in Arm A will be treated with combination pembrolizumab and carboplatin followed by maintenance pembrolizumab if stable or responding disease.

Participants in Arm B will be treated with carboplatin only until disease progression, whereupon they may crossover to receive pembrolizumab with or without carboplatin at investigator's discretion (Arm Bx). After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events will be collected for 90 days after the end of treatment. Participants who discontinue for reasons other than progressive disease will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent, becoming lost to follow-up, or death.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced breast cancer with locally recurrent chest wall disease not amenable to surgical excision with curative intent.

   1. Distant sites of disease are allowed
   2. Prior radiation to the chest wall is not required
2. The following disease subtypes are eligible:

   1. Triple negative disease (defined as ER < 10%, PR < 10%, HER2 negative)
   2. Hormone receptor positive, HER2 negative disease with evidence of progression on at least two prior lines of hormone therapy, unless, per treating investigator's judgement, is not considered a candidate for further endocrine therapy
   3. HER2 positive disease with evidence of disease progression on trastuzumab, pertuzumab, Trastuzumab emtansine (T-DM1), and oral tyrosine kinase inhibitor unless contraindicated with no other HER2 targeted therapy options available. Patients in this category will be classified by ER status

      * Histologically confirmed HER2+ breast carcinoma, with HER2+ defined by in situ hybridization (ISH) or fluorescence in situ hybridization (FISH) or immunohistochemistry (IHC) methodology using standard criteria.
      * Cardiac function must be determined within 4 weeks of study entry to be >= institutional lower limit of normal (LLN) using echo or multiple gated acquisition scan (MUGA).
3. Any number of prior lines of therapy are allowed. a Prior platinum based therapy is allowed in the following settings:

   * Treatment in the neoadjuvant and/or adjuvant setting without clear progression of disease.
   * Treatment in the metastatic setting without clear progression of disease. b Neo/adjuvant treatment with a checkpoint inhibitor is allowed if the last treatment was at least 12 months from the diagnosis of metastatic disease.
4. At least two weeks from last systemic therapy for breast cancer, with recovery of all treatment related toxicity to grade 1 or less. Subjects with <= Grade 2 neuropathy are an exception to this criterion.
5. At least two weeks from last radiation therapy, with recovery of all treatment related toxicity to grade 1 or less (excluding alopecia).
6. Prior CNS disease is allowed if stable for at least one month since whole brain radiation therapy, and 2 weeks since stereotactic radiotherapy, and not requiring steroids. Patients whose CNS disease was surgically treated may be enrolled if stable for at least one month, and not requiring steroids.
7. Able to provide tissue from a newly obtained core or excisional biopsy of a chest wall tumor lesion. Newly-obtained is defined as a specimen any time after the last systemic or local therapy utilized to treat the disease. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
8. Willing and able to provide written informed consent.
9. Greater than or equal to 18 years of age on day of signing informed consent.
10. Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2.
11. Adequate organ function as defined below within 10 business days of treatment initiation:

    * Absolute neutrophil count (ANC) >=1,000 /microliter (mcL)
    * Platelets>=100,000 / mcL
    * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
    * Serum creatinine OR Measured or calculated* creatinine clearance (GFR can also be used in place of creatinine or CrCl) <=1.5 X upper limit of normal (ULN) OR >=60 mL/min for subject with creatinine levels > 1.5 X institutional ULN. Creatinine clearance should be calculated per institutional standard.
    * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin <= ULN for subjects with total bilirubin levels > 1.5 ULN
    * Aspartate aminotransferase (AST) (SGOT) and Alanine aminotransferase (ALT) (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
    * Albumin >2.5 g/dL
    * International Normalized Ratio (INR) or Prothrombin Time (PT) <=1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    * Activated Partial Thromboplastin Time (aPTT) <=1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
12. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential should be willing to use an acceptable form of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
14. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Treatment with an investigational agent within 4 weeks of the first dose of treatment.
2. A diagnosis of immunodeficiency or is currently receiving systemic steroid therapy at any dose or is receiving any other form of immunosuppressive therapy. Steroid therapy is not allowed within 7 days prior to the first dose of trial treatment. However, topical and intranasal corticosteroids are allowed, and not an exclusion for participation.
3. Known active TB (Bacillus Tuberculosis). Patients with a distant history of tuberculosis that was appropriately treated and have no evidence of active infection are eligible to participate. Patients with a history of latent tuberculosis that was appropriately treated are also eligible to participate.
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Hypersensitivity to carboplatin or cisplatin
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/ interstitial lung disease
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Prior checkpoint inhibitor therapy in the metastatic setting.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B virus (HBV) [e.g., hepatitis B surface antigen (HBsAg) reactive] or Hepatitis C virus (HCV) [e.g., HCV ribonucleic acid (RNA), [qualitative] is detected].
18. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Huppert, MD, BA, Principal Investigator — University of California, San Francisco; Neelima Vidula, MD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - University of California, San Francisco, San Francisco, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Background] Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, Jungbluth A, Gnjatic S, Thompson JA, Yee C. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med. 2008 Jun 19;358(25):2698-703. doi: 10.1056/NEJMoa0800251. PMID 18565862
- [Background] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Background] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, Qiu Y, Jussif JM, Carter LL, Wood CR, Chaudhary D. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004 Sep 10;574(1-3):37-41. doi: 10.1016/j.febslet.2004.07.083. PMID 15358536
- [Background] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Pembrolizumab + Carboplatin: Participants receive carboplatin intravenously (IV) and pembrolizumab IV over 30 minutes on day 1. Participants who are human epidermal growth factor receptor 2 positive (HER2+) also receive trastuzumab IV every 3 weeks. Treatment repeats every 3 weeks for a least 6 courses in the absence of disease progression or unacceptable toxicity. After completion of 6 cycles of carboplatin and pembrolizumab, participants with stable or responding disease receive pembrolizumab monotherapy on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
- Arm B: Carboplatin Monotherapy, then Pembrolizumab for participants who progress only: Participants receive carboplatin on day 1. Patients who are HER2+ also receive trastuzumab IV every 3 weeks. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Participants with disease progression (PD) are eligible to receive pembrolizumab on day 1 of each cycle (crossover). Carboplatin may be continued or added back into the treatment regimen at the investigator's discretion. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
Period: Treatment assigned at enrollment
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy, then Pembrolizumab for participants who progress only
Started | 52 | 24
Completed | 51 | 24
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Patients who Progressed on Arm B
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy, then Pembrolizumab for participants who progress only
Started (Arm A participants not eligible for crossover) | 0 | 16
Completed | 0 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy | Total
Number analyzed (Participants) | 52 | 24 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.19 (12.11) | 59.62 (11.22) | 56.59 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 24 | 76
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 47 | 18 | 65
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 4 | 7
  White | 39 | 13 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 52 | 24 | 76

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) at 18 Weeks
Description: The percentage of participants with Complete response (CR), Partial Response (PR), and stable disease (SD) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at 18 weeks of treatment in breast cancer patients with chest wall disease treated with pembrolizumab and carboplatin (Arm A) or carboplatin alone (Arm B) will be reported.
Time Frame: Up to 18 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy, then Pembrolizumab for participants who progress only
Number analyzed (Participants) | 51 | 24
percentage of participants | 20 | 17

2. Primary Outcome: Median Progression Free Survival (PFS) at 18 Weeks
Description: PFS is defined as the time in months from observed objective response to disease progression at week 18 and will be summarized using estimates by the Kaplan-Meier method in order to account for any censoring participants by enrolling treatment arms (Arm A and Arm B only)
Time Frame: Up to 18 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy
Number analyzed (Participants) | 51 | 24
months | 2.06 [1.38 to 3.12] | 2.63 [1.44 to 4.17]

3. Secondary Outcome: DCR by Immune-related (ir) RECIST at 18 Weeks
Description: The percentage of participants with Complete response (CR), Partial Response (PR), and stable disease (SD) as defined by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) at 18 weeks of treatment in breast cancer patients with chest wall disease treated with pembrolizumab and carboplatin (Arm A) or carboplatin alone (Arm B) and also based on PD-L1 expression
Time Frame: Up to 18 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy
Number analyzed (Participants) | 51 | 24
percentage of participants | 18 | 17

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR will be presented as the percentage of participants with CR or PR as determined by RECIST criteria.
Time Frame: Up to 18 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy
Number analyzed (Participants) | 51 | 24
percentage of participants | 8 | 12.5

5. Secondary Outcome: Number of Participants With Treatment-related Adverse Events (AEs)
Description: Adverse events will be graded and recorded according to NCI CTCAE Version 4.0 up to 30 days after the last treatment. Grade 1 laboratory abnormalities and white blood cell differential abnormalities excluding neutrophils (i.e., lymphocytes, monocytes, basophils, etc.) did not need to be recorded as adverse events.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm BX: Arm B Participants Who Progressed: Participants with disease progression (PD) are eligible to receive pembrolizumab on day 1 of each cycle (crossover). Carboplatin may be continued or added back into the treatment regimen at the investigator's discretion. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Participants who are HER2+ also receive trastuzumab IV every 3 weeks.
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy | Arm BX: Arm B Participants Who Progressed
Number analyzed (Participants) | 51 | 24 | 16
Participants | 33 | 12 | 6

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: Per protocol, Grade 1 laboratory abnormalities and white blood cell differential abnormalities excluding neutrophils (i.e., lymphocytes, monocytes, basophils, etc.) were not recorded as AEs.
Groups:
- Arm BX: Participants who progressed on Arm B: Participants with disease progression (PD) are eligible to receive pembrolizumab on day 1 of each cycle (crossover). Carboplatin may be continued or added back into the treatment regimen at the investigator's discretion. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Participants who are HER2+ also receive trastuzumab IV every 3 weeks.
Arm/Group | Arm A: Pembrolizumab + Carboplatin | Arm B: Carboplatin Monotherapy | Arm BX: Participants who progressed on Arm B
All-Cause Mortality (participants affected / at risk) | 15/52 | 2/24 | 4/16
Serious Adverse Events (participants affected / at risk) | 15/52 | 2/24 | 4/16
Other Adverse Events (participants affected / at risk) | 43/52 | 19/24 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pembrolizumab + Carboplatin (N=52) | Arm B: Carboplatin Monotherapy (N=24) | Arm BX: Participants who progressed on Arm B (N=16)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Febrile Neurtopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspenea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pembrolizumab + Carboplatin (N=52) | Arm B: Carboplatin Monotherapy (N=24) | Arm BX: Participants who progressed on Arm B (N=16)
Anemia (Blood and lymphatic system disorders) | 14 (29) | 4 (10) | 1 (2)
Blood and Lymphatic System Disorders - Other, specify (Blood and lymphatic system disorders) | 5 (12) | 2 (2) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 13 (15) | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Breast infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 9 (15) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 18 (35) | 4 (6) | 2 (4)
Platelet count decreased (Investigations) | 16 (31) | 4 (5) | 3 (3)
White blood cell decreased (Investigations) | 10 (18) | 2 (2) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (14) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 5 (10) | 2 (4)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/52/NCT03095352/Prot_SAP_000.pdf